CLINICAL TRIAL: NCT03614026
Title: Randomized Controlled Trial of Teachers and Parents as Partners During Middle School
Brief Title: Teachers and Parents as Partners During Middle School RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0165; A173000 (Other: UW Madison); EDUC/EDUC PSYCHOLOGY (Other: UW Madison); R324B160043 (Other Grant/Funding Number: US Dept of Education); Protocol Version 7/29/2020 (Other: UW Madison)
Record Dates: First submitted 2018-07-22; First posted 2018-08-03 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Behavior Disorders
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: Intervention condition and business-as-usual control condition
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teachers and Parents as Partners Intervention (Experimental): Teachers and Parents as Partners will occur in a series of stages comprised of approximately four structured meetings over approximately 8 weeks. A Teachers and Parents as Partners consultant will meet together with a student's parent(s), teachers, other school personnel (as appropriate), and the student (as appropriate). The Teachers and Parents as Partners team will collaboratively address behavior problem solving objectives. Specific objectives include: identifying strengths and specific behaviors of concern, specifying alternative prosocial behaviors, creating measurable behavior goals, co-constructing behavior intervention/support plans to address the target concerns, creating sustainable conditions to support plan implementation at home and school, and evaluating the plan to assess progress toward goals.
  Interventions: Behavioral: Teachers and Parents as Partners
- Business as usual control (No Intervention): In the business-as-usual control condition, participants will have access to any services that a school would routinely provide (e.g., develop and implement a behavior support plan) as well as services families can access in the community (e.g., mental health support).

INTERVENTIONS:
Behavioral: Teachers and Parents as Partners — Family-school partnership intervention
  Arms: Teachers and Parents as Partners Intervention

SUMMARY:
There are two aims of this study (a) to examine the effect of Teachers and Parents as Partners on student, parent, and teacher outcomes in middle school and (b) identify barriers and facilitators to implementing Teachers and Parents as Partners in middle school for students with behavior concerns.

DETAILED DESCRIPTION:
In the business-as-usual control condition, participants will have access to any services that a school would routinely provide (e.g., develop and implement a behavior support plan) as well as services families can access in the community (e.g., mental health support).

Teachers and Parents as Partners will occur in a series of stages comprised of approximately four structured meetings over approximately 8 weeks. A Teachers and Parents as Partners consultant will meet together with a student's parent(s), teachers, other school personnel (as appropriate), and the student (as appropriate). The Teachers and Parents as Partners team will collaboratively address behavior problem solving objectives. Specific TAPP objectives include: identifying strengths and specific behaviors of concern, specifying alternative prosocial behaviors, creating measurable behavior goals, co-constructing behavior intervention/support plans to address the target concerns, creating sustainable conditions to support plan implementation at home and school, and evaluating the plan to assess progress toward goals.

ELIGIBILITY:
Inclusion Criteria:

* Students will be eligible if they have scores in the "elevated" or "extremely elevated" risk categories on the parent or teacher version of the Behavior Assessment Scale for Children (BASC) 3 Behavioral and Emotional Screening System (BESS). Parents, and primary teachers and school staff associated with an eligible student will be included.

Exclusion Criteria:

* Students who do not meet the inclusion criteria will be excluded from participation, which includes their parent(s), teachers, and other school personnel. Students also may not be eligible if they have mental health concerns or severe behavior problems that may not be appropriate for Teachers and Parents as Partners or a research project (e.g., some internalizing problems, students who pose an risk of harming themselves).

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2018-09-30 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Behavior Assessment Scale for Children (assessing change) | pretest and about 12 weeks later at posttest
  Report of child behavior
Social Skills Improvement System (assessing change) | pretest and about 12 weeks later at posttest
  Report of child social skills
Direct behavior rating (assessing change) | Time series during the approx 12 week intervention
  Ratings of child behavior
Goal attainment scaling (through study completion) | At the conclusion of the intervention
  Ratings of goals met

SECONDARY OUTCOMES:
Academic Competence Evaluation (assessing change) | pretest and about 12 weeks later at posttest
  Reports of child academic competence
Parent-teacher relationship scale (assessing change) | pretest and about 12 weeks later at posttest
  Ratings of the parent-teacher relationship
Competence in problem solving (assessing change) | pretest and about 12 weeks later at posttest
  Parent and teacher ratings of their competence in problem solving
Parent monitoring scale (assessing change) | pretest and about 12 weeks later at posttest
  Ratings of parent monitoring child activities
Behavior intervention rating scale-revised (through study completion) | At the conclusion of the intervention
  Ratings of intervention acceptability
Work completion (assessing change) | Time series during the approx 12 week intervention
  Ratings of student work completion

CONTACTS AND LOCATIONS:
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Undecided
This study is funded by the Institute of Education Sciences. Thus, we comply with the IES policy on data sharing as well as other policies and regulations governing research awards.